CLINICAL TRIAL: NCT04760327
Title: Electrochemotherapy of Gynecological Cancers
Acronym: GynECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0120-692/2017/4
Record Dates: First submitted 2018-04-05; First posted 2021-02-18 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Gynecological Cancers
Keywords: Electrochemotherapy; Cisplatin; Bleomycin
MeSH Terms: interventions — Electrochemotherapy; Bleomycin; Cisplatin; Electroporation; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrochemotherapy of gynecological cancers (Experimental)
  Interventions: Combination Product: Electrochemotherapy with bleomycin or cisplatin

INTERVENTIONS:
Combination Product: Electrochemotherapy with bleomycin or cisplatin — Electrochemotherapy with cisplatin or bleomycin of gynecological cancers
  Other Names: Combination of drug delivery platform (electroporation) and drug (bleomycin or cisplatin)

SUMMARY:
To determine the effectiveness, feasibility and safety of electrochemotherapy in treatment of local and/or regional recurrences of gynecological cancers with electrochemotherapy in which standard treatment options have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

1. Local or regional relapse of gynecological tumors in which standard treatment options have been exhausted.
2. Age more than 18.
3. Life expectancy more than 3 month.
4. Performance status Karnofsky ≥ 70 or WHO < or 2.
5. Treatment free interval minimum 2 weeks.
6. Patient must be mentally capable of understanding the given information and regarding treatment and any adverse reactions that may occur during treatment.
7. Patient must give informed consent.
8. Patient must be discussed at the multidisciplinary team before entering the trial.
9. Patient should be suitable for anesthesia.

Exclusion Criteria:

1. Visceral, bone or diffuse metastases.
2. Life-threatening infection and/or heart failure and/or liver failure and/or other severe systemic pathologies.
3. Significant reduction in respiratory function.
4. Age less than 18 years.
5. Coagulation disturbances (those who do not respond on standard treatment with vitamin-K or fresh frozen plasma).
6. Cumulative dose of ≥ 400 mg/m2 bleomycin received.
7. Impaired kidney function (creatinin > 150 µmol/l).
8. Patients with epilepsy.
9. Pregnancy.
10. Patient incapable of understanding the aim of the study or disagree with the entering into the clinical study.

Ages: 18 Years to 105 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of electrochemotherapy according to RECIST 1.1 criteria. | Changes from baseline regularly up to 24 months
  Effectiveness of electrochemotherapy in the treatment of local or regional recurrences of gynecological tumors in which standard treatment options have been exhausted. Effectiveness will be evaluated according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Safety of electrochemotherapy according to CTCAE v5.0 criteria. | during hospitalization and up to 24 months
  To determine safety of electrochemotherapy in the treatment of local or regional recurrences of gynecological tumors in which standard treatment options have been exhausted. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 criteria will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of oncology Ljubljna, Ljubljana, Slovenia